CLINICAL TRIAL: NCT02889588
Title: Visual and Optics Impact of Refractive Surgery
Acronym: CRIVO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DGL_2015_20
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Refractive Disorders
Keywords: Refractive Surgery; higher order aberrations
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Refractive surgery includes interventions to correct refractive errors, using a medical device such as a laser or an implant (intraocular lenses) or surgical instruments. The study distinguishes corneal interventions, carried on the surface of the eye, and intraocular interventions, performed on the lens or in the anterior or posterior chamber of the eye. The number of procedures in refractive surgery is growing significantly. They seem to offer satisfactory visual results but a number of issues remains unresolved. In order to get emmetropia, refractive surgery corrects optical defects by decreasing aberrations of lower orders (ie spherical refractive error and astigmatism). This increases high-order aberrations (the most common is a bright halo on the edge of the image). The cutting of the flap to the surface of the cornea in the case of LASIK increases high-order aberrations, which have the effect of reducing post-surgical visual performance (ie visual acuity and contrast sensitivity) and can't be corrected by glasses, while the adaptation of contact lenses on a post-operative cornea is more complex. It is therefore necessary to limit these post-surgical aberrations and to identify their possible sources. Indeed, some authors have provided insight into the effects of some high-order aberrations, but the influence of several factors characterizing the preoperative eye on refractive surgery are still unknown, such as pupillary diameter, depth of the anterior chamber, Intra Ocular Pressure or astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* patient candidate for Laser in Situ Keratomileusis (LASIK) refractive surgery
* 18 to 40 years old
* corrective glasses or lenses ranging from -9.00 to + 6.00 diopter
* astigmatism less than or equal to 5 diopter

Exclusion Criteria:

* patient opposition to participate in the study
* patient under legal protection
* Pregnant or breast feeding patient
* no health insurance coverage

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing refractive surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
number of high order aberrations after refractive surgery | 3 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Imène SALAH, Study Director — Fondation OPH A de Rothschild; Damien GATINEL, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France